CLINICAL TRIAL: NCT01521156
Title: Cholesterol Lowering Effects of a Drinkable Low Fat Dairy Product Enriched With Plant Sterols
Brief Title: Effect of the Consumption of a Fermented Dairy Product Enriched With Plant Sterols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NU312
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Mild Hypercholesterolemic Subjects
Keywords: Plant sterols - Hypercholesterolemia - Diet - Dairy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Control product (Active Comparator)
  Interventions: Other: 1- low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols).
- 2 = Tested product (Experimental)
  Interventions: Other: 2- low-fat dairy fermented product (drinkable) enriched with experimental plant sterols-esters (1,6g /day equivalent as free sterols).

INTERVENTIONS:
Other: 1- low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols). — 1 = Intervention 1 (1 test product/day)
  Arms: 1 = Control product
Other: 2- low-fat dairy fermented product (drinkable) enriched with experimental plant sterols-esters (1,6g /day equivalent as free sterols). — 2 = Intervention 2 (1 test product/day)
  Arms: 2 = Tested product

SUMMARY:
The purpose of this study is to investigate the cholesterol lowering effect of a drinkable low fat fermented milk enriched with plant sterols after 3 weeks of daily consumption in midly hypercholesterolemic people.

ELIGIBILITY:
Inclusion Criteria:

* Male/female subject, aged from 18 to 75,with BMI between 18,5 and 30 kg/m², with LDL-cholesterol blood level between 130 mg/dL to 190 mg/dL without statin therapy.
* Subject accepting to follow the dietary recommendations advisable for hypercholesterolemic subject.
* Subject used to consume dairy products.
* For female subjects: effective contraceptive methods used.
* Subject having given written consent to take part in the study.

Exclusion Criteria:

* Subject with blood triglycerides levels above 350 mg/dL.
* Subject having experienced any cardiovascular event in the last 6 months.
* Subject having sitosterolemia.
* Subject taking any hypocholesterolemic treatment drugs.
* Intake of blood lipid-regulating supplementation of blood lipid-regulating dietary supplements or functional food during the last 2 weeks before study start.
* Diabetic subject (type I and type II).
* Subject smoking strictly more than 10 cigarettes / day.
* Subject with heavy alcohol intake (> 40 g / day for men ; > 30 g / day for women).
* Subject presenting known allergy or hypersensitivity to milk proteins.Subject with known soy allergy.
* Subject refusing to stop the consumption of plant sterols-enriched products if any during the study (other than the studied product).
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters.
* Subject receiving a transplant and under immunosuppressor treatment.
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial.
* Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.
* Subject with any kind of disease likely to interfere with the evaluation of efficiency or safety of the product.
* For female subject: pregnancy, breast feeding or intention to be pregnant during the study.
* For female subject: subject likely to change her contraceptive method during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harrison Clinical Research Clinical Unit, Munich, Germany